CLINICAL TRIAL: NCT04005248
Title: Prevalence of Undiagnosed HCV Infections in HIV-negative MSM Visiting a Sexual Health Clinic.
Brief Title: Prevalence of HCV in HIV-negative MSM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: Public Health Service of Rotterdam-Rijnmond (Unknown)
Responsible Party: Principal Investigator, Bart Rijnders, Principal Investigator, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MEC-2019-0105; IN-NL-987-4652 (Other Grant/Funding Number: Gilead Sciences)
Record Dates: First submitted 2019-06-25; First posted 2019-07-02 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Intervention Model Description: Cross-sectional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Testing for HCV (Other): HCV IgG test and questionnaire; both at visit to the sexual health clinic
  Interventions: Diagnostic Test: HCV IgG test

INTERVENTIONS:
Diagnostic Test: HCV IgG test — An HCV IgG test (performed on blood already collected for regular STI tests), combined with a questionnaire on sexual risk behavior. If client is HCV IgG positive, a HCV RNA test will be performed.

SUMMARY:
This study measures the prevalence of undiagnosed hepatitis C virus (HCV) infection in HIV-negative men-who-have-sex-with-men (MSM) visiting the sexual health clinics of public health services (in dutch: gemeentelijke gezondheidsdienst, GGD), in order to evaluate if systematic screening for HCV of HIV-negative MSM attending sexual health clinics in the Netherlands is needed.

DETAILED DESCRIPTION:
Until recently, sexually acquired HCV infections were thought to be limited to HIV-positive MSM. Yet, emerging data show that the prevalence of HCV among HIV uninfected MSM that opt-in for HIV pre-exposure prophylaxis (PrEP) is much higher. It was 5% (n=18/375) in Amsterdam and 2% (n=4/200) in Antwerp (Be-PrEP-ared; EudraCT2015-000054-37) (23).

This observation may be the result of the fact that PrEP users are, by definition, at risk for sexually transmitted infections because PrEP is only prescribed to those at risk for HIV. However, another explanation may be that in the new context of HIV "treatment as prevention" and the availability of PREP as a way to protect oneself against HIV, the incidence of HCV in HIV uninfected MSM is changing. Furthermore, if PrEP use would lead to an increase in sexual risk-taking, this may eventually lead to an increase in the incidence of HCV among HIV negative MSM on PrEP. If these HCV infections among HIV negative MSM remain unnoticed, they are a continuous source of HCV infections in HIV+MSM as well for the larger HIV-MSM community. Furthermore, PrEP as well as the very well-documented efficacy of HIV treatment as prevention can be expected to increase sexual mixing of HIV- and HIV+MSM.

Based on the observations described above, we hypothesize that undiagnosed HCV infections in HIV negative MSM are (or may become) an important source of HCV (re)infections in HIV+MSM as well as the larger HIV-MSM population.

Primary objectives:

1. Measure the prevalence of HCV in a large group of HIV-negative MSM attending sexual health clinics in the Netherlands.
2. Assess Risk Factors for HCV in order to validate the HCV-MOSAIC risk score in HIV-MSM, which may allow for a more cost-effective (=targeted) HCV testing of HIV-MSM in the future

Secondary objectives:

1. Measure the acceptability of HCV testing in HIV-MSM at public health clinics.
2. Evaluate the HCV outcome in terms of the proportion of HCV infections that cleared spontaneously (= HCV IgG positive but HCV RNA negative) versus the total number of HCV IgG positive clients.

The HCV-immunoglobulin G (IgG) test is offered on top of the regular sexually transmitted infection (STI) tests. A positive HCV-IgG test will be followed by an HCV-RNA test. Clients known to be HCV IgG positive as a result of a previous HCV infection will be tested for HCV using an HCV-RNA test.

Before HCV testing, participants will be asked to fill out a detailed study questionnaire about possible risk factors for HCV acquisition (PREP use, receptive unprotected anal intercourse, use of non-IV or injection drugs during sex, fisting, recent diagnosis of ulcerative rectal STI, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Self-identifying as a man-who-has-sex-with-men (MSM)
* Willing to undergo HCV testing

Exclusion Criteria:

* Clients known to be HIV positive

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
HCV antibody prevalence | From start study to end of study, at least 2 years
  Percentage of HCV IgG antibody positive clients per 1000 HIV-negative MSM tested
Value of HCV-MOSAIC risk score in HIV-negative MSM | From start study to end of study, at least 2 years
  Assess risk factors for a positive HCV IgG test in the study population according to the HCV-MOSAIC risk score, using sexual behavior questionnaires. The HCV-MOSAIC risk score is validated to identify HIV+MSM at risk for an acute HCV infection (Newsum et al, 2017).
  HCV-MOSAIC risk score:
  * Condomless receptive anal intercourse in the last 6 months - 1.1
  * Sharing of sex toys in the last 6 months - 1.2
  * Unprotected fisting in the last 6 months - 0.9
  * Injecting drug use in the last 12 months - 1.4
  * Sharing of straws when using nasally administered drug in the last 12 months - 1.0
  * Ulcerative STI in the last 12 months - 1.4
  Cut-off sum ≥2.0 = at risk for acute HCV infection

SECONDARY OUTCOMES:
HCV infection prevalence | From start study to end of study, at least 2 years
  Prevalence of active HCV infection (RNA positive) among those with HCV IgG antibodies
Proportion participating in study | From start inclusion to end of inclusion period, at least 1 year
  Percentage of HIV-negative MSM that accepted to be tested for HCV

CONTACTS AND LOCATIONS:
Overall Officials: Bart J.A. Rijnders, MD PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- GGD Rotterdam Rijnmond, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoornenborg E, Achterbergh RCA, Schim van der Loeff MF, Davidovich U, Hogewoning A, de Vries HJC, Schinkel J, Prins M, van de Laar TJW; Amsterdam PrEP Project team in the HIV Transmission Elimination AMsterdam Initiative, MOSAIC study group. MSM starting preexposure prophylaxis are at risk of hepatitis C virus infection. AIDS. 2017 Jul 17;31(11):1603-1610. doi: 10.1097/QAD.0000000000001522. PMID 28657964
- [Background] Vanhommerig JW, Lambers FA, Schinkel J, Geskus RB, Arends JE, van de Laar TJ, Lauw FN, Brinkman K, Gras L, Rijnders BJ, van der Meer JT, Prins M; MOSAIC (MSM Observational Study of Acute Infection With Hepatitis C) Study Group; van der Meer JT, Molenkamp R, Mutschelknauss M, Nobel HE, Reesink HW, Schinkel J, van der Valk M, van den Berk GE, Brinkman K, Kwa D, van der Meche N, Toonen A, Vos D, van Broekhuizen M, Lauw FN, Mulder JW, Arends JE, van Kessel A, de Kroon I, Boonstra A, van der Ende ME, Hullegie S, Rijnders BJ, van de Laar TJ, Gras L, Smit C, Lambers FA, Prins M, Vanhommerig JW, van der Veldt W. Risk Factors for Sexual Transmission of Hepatitis C Virus Among Human Immunodeficiency Virus-Infected Men Who Have Sex With Men: A Case-Control Study. Open Forum Infect Dis. 2015 Aug 6;2(3):ofv115. doi: 10.1093/ofid/ofv115. eCollection 2015 Sep. PMID 26634219
- [Background] Newsum AM, Stolte IG, van der Meer JT, Schinkel J, van der Valk M, Vanhommerig JW, Buve A, Danta M, Hogewoning A, Prins M; MOSAIC collaborators. Development and validation of the HCV-MOSAIC risk score to assist testing for acute hepatitis C virus (HCV) infection in HIV-infected men who have sex with men (MSM). Euro Surveill. 2017 May 25;22(21):30540. doi: 10.2807/1560-7917.ES.2017.22.21.30540. PMID 28597832